CLINICAL TRIAL: NCT04872413
Title: A Pilot Study of Interrogating Biological Signaling Pathway Dysregulations and In Vitro Screening With Personalized Therapies in Resistant Mantle Cell Lymphoma (MCL) - the MCL MATCH Trial
Brief Title: Interrogating Biological Signaling Pathway Dysregulations and In Vitro Screening With Personalized Therapies in Relapsed or Refractory Mantle Cell Lymphoma, MCL MATCH Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-1022; NCI-2021-02576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1022 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Chromatin Immunoprecipitation Sequencing; Follow-Up Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (biospecimen collection) (Experimental): Patients undergo blood, saliva or tissue sample collection for mRNA analysis and drug efficacy testing. Patients assigned treatment per the results are followed every 1 cycle of therapy for 1 year, every 2 months for 1 year, every 4 months for 1 year then every 6 months thereafter.
  Interventions: Procedure: Biospecimen Collection; Other: Follow-Up

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood, saliva or tissue sample collection
Other: Follow-Up — Undergo follow-up
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup

SUMMARY:
This clinical trial collects and tests samples using genetic testing to find personalized treatments that may work best for patients with mantle cell lymphoma (MCL) that has come back (relapsed) or does not respond to treatment (refractory). Several types of MCL are difficult to treat due to specific genetic changes (mutations or alterations in the DNA/RNA expression in the cells) that make them not respond to a certain type of drug called a Bruton's tyrosine kinase (BTK) inhibitor. The goal of this clinical research study is to use genetic testing to identify which drugs may be most effective in treating patients with MCL who have this type of genetic mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of the proposed therapy based on dysregulated cell signaling pathways in combination with in vitro drug activity.

SECONDARY OBJECTIVES:

I. Overall response rates (complete response [CR] + partial response [PR]). II. Safety in patients who were treated with matched personalized therapies. III. Duration of response. IV. Progression free survival (PFS). V. Overall survival (OS).

EXPLORATORY OBJECTIVE:

I. Correlation of somatic mutations in MCL with cell signaling dysregulated activity and therapeutic implications of somatic mutations in relapsed MCL.

OUTLINE:

Patients undergo blood, saliva or tissue sample collection for messenger ribonucleic acid analysis (mRNA) analysis and drug efficacy testing. Patients assigned treatment per the results are followed every 1 cycle of therapy for 1 year, every 2 months for 1 year, every 4 months for 1 year then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed MCL tissue diagnosis with CD20- and Cyclin D1-positive cells or cyclin D1 negative but t (11;14) positive and diagnosis confirmed by pathologist from the tissue biopsy.
2. Patients must have relapsed/refractory MCL.
3. Understand and voluntarily sign an IRB-approved informed consent form.
4. Patients must have a biopsy-accessible lesion and be willing to undergo biopsy.
5. Patients must have bi-dimensional measurable disease per Cheson criteria (bone marrow or GI-only involvement is acceptable).
6. Age ≥ 18 years at the time of signing the informed consent.
7. Absolute neutrophil count ≥ 1.0 x 109/L, absolute lymphocyte count ≥ 0.6 x 109/L, platelet count ≥ 50 x 109/L
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
9. Patients must have adequate organ function for drugs(s) or combination being utilized (dependent on the drug (s) being given, the acceptable values of clinical parameters are given below: Biochemical values should be within the following limits:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
   3. Creatinine clearance (CLcr) > 30 mL/min
10. Cardiac ejection fraction ≥ 50% by ECHO or MUGA.
11. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test. Men must agree not to father a child and agree to use a condom if his partner is of child-bearing potential.

Exclusion Criteria:

1. Any serious medical condition that places the patient at unacceptable risk and/or would prevent the subject from signing the informed consent form. Examples include but are not limited to uncontrolled hypertension, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, active infection, active hemorrhage, and psychiatric illness.
2. Patient with rapid progressive disease, warranting urgent immediate admission.
3. Pregnant or breastfeeding females.
4. Known HIV infection or active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum Hepatitis B antibody). Known hepatitis C infection is allowed as long as there is no active disease and is cleared by GI-Hepatology consultation.
5. The patient has a prior or concurrent malignancy that, in the opinion of the investigator, presents a greater risk to the patient's health and survival than the MCL, with a life expectancy ≤ 1 year.
6. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure or myocardial infarction within 6 months at the time of consent, or any cardiac disease defined by the New York Heart Association Classification as Class 3 (moderate) or 4 (severe).
7. Prior chemotherapy within 2 weeks, nitrosoureas within 6 weeks, therapeutic anticancer antibodies within 2 weeks, radio- or toxin-immunoconjugates within 2 weeks, radiation therapy or other investigational agents within 1 week, major surgery within 4 weeks, or vaccination with live attenuated vaccines within 4 weeks of the first dose of start of assigned therapy.
8. The patient receives corticosteroids for non-malignant conditions (e.g., asthma, inflammatory bowel disease) equivalent to a dexamethasone dose ≥ 4 mg/day or prednisone ≥ 20 mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Feasibility rate | Up to 1 year
  Will be reported by frequency with exact 95% confidence interval. Logistic regression will be utilized to assess the effect of patient prognostic factors on the feasibility and response rate.

SECONDARY OUTCOMES:
Response rate | Up to 1 year
  Will be reported by frequency with exact 95% confidence interval. Logistic regression will be utilized to assess the effect of patient prognostic factors on the feasibility and response rate.
Incidence of adverse events | Up to 1 year
  Toxicity data by type and severity will be summarized by frequency tables.
Duration of response | Up to 1 year
Progression free survival | Up to 1 year
  Will be estimated using the method of Kaplan and Meier. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.
Overall survival | Up to 1 year
  Will be estimated using the method of Kaplan and Meier. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.

OTHER OUTCOMES:
Correlation of somatic mutations in mantle cell lymphoma with cell signaling dysregulated activity | Up to 1 year
  Will be estimated using the method of Kaplan and Meier. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT04872413/ICF_000.pdf